CLINICAL TRIAL: NCT01388075
Title: Genetic Variability in the Response to Warfarin at Baseline and During Induction of CYP2C9
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Mordechai Muszkat, MD, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: HMO-0451-10
Record Dates: First submitted 2011-07-03; First posted 2011-07-06 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Healthy Subjects
Keywords: induction; CYP2C9; Genetic variability; Expression
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rifampicin (Experimental): Consecutive treatments with rifampicin and placebo
  Interventions: Drug: Rifampicin

INTERVENTIONS:
Drug: Rifampicin — oral, 450 mg/day , 7 days

SUMMARY:
The genetic factors associated with variability in CYP2C9 induction have not been elucidated. The hypothesis underlying this study is that following 7 days treatment with rifampicin, a known CYP450 inducer, the genetic variability in regulatory elements controlling CYP2C9 expression will be associated with the magnitude of change in INR response to warfarin and in CYP2C9-mediated warfarin metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Consumption of any medication during 30 days
* Smoking
* Alcohol consumption

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-07; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
International Normalized Ratio (INR) | 6 weeks

SECONDARY OUTCOMES:
Warfarin concentration | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel